CLINICAL TRIAL: NCT07330544
Title: A Phase II Clinical Study Evaluating Entinostatwit h or Without Anlotinib + Fulvestrant for the Treatment of Hormone Receptor (HR) -Positive, Human Epidermal Growth Factor Receptor-2 (HER-2) -Negative Advanced Breast Cancer That Relapsed or Progressed After Endocrine Therapy
Brief Title: A Phase II Clinical Study Evaluating Entinostat With or Without Anlotinib + Fulvestrant for the Treatment of Hormone Receptor (HR) -Positive, Human Epidermal Growth Factor Receptor-2 (HER-2) -Negative Advanced Breast Cancer That Relapsed or Progressed After Endocrine Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Hu Hai, Chief of Breast Internal Medicine Department, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAF-BC-IIT-001
Record Dates: First submitted 2025-11-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat; Fulvestrant; anlotinib

STUDY DESIGN:
Intervention Model Description: The study adopted the Simon phase 2 design, and all 20 eligible patients were treated with entinostat + fulvestrant; The study was terminated if no more than 2 patients achieved objective response and continued to enter Phase 2 if no more than 3 patients achieved objective response. In Phase 2, qualified patients were randomly assigned at a ratio of 1:1.5 to either the entinostat + fluvestrant group (Group 1) or the anlotinib + entinostat + fluvestrant group (Group 2), with 39 patients enrolled in group 1 and 59 patients enrolled in group 2; All patients were treated until the subjects' treatment would continue until the subjects experienced disease progression, intolerable toxicity, active withdrawal from treatment, or other conditions specified in the protocol, whichever occurred first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- entinostat + fulvestrant (Experimental): Entinostat tablets Dosage form: Tablets Specification Appearance: 1.0 mg (pink to pale red) or 5.0 mg/ tablet (yellow) Dosage and Administration: 1 tablet (5 mg/ tablet) once a week, orally administered. Take at least 1 hour before meals or at least 2 hours after meals.
  Combination therapy:
  Fulvestrant injection Dosage form: Injection Appearance: A clear, viscous, colorless to yellowish liquid Specification: 5 ml; 0.25g per vial Dosage and Administration: 500 mg by intramuscular injection. Each 28-day treatment cycle is administered on day 1 and day 15 of the first cycle, followed by day 1 of each subsequent cycle
  Interventions: Drug: entinostat; Drug: Fulvestrant
- entinostat + fulvestrant+anlotinib (Experimental): Entinostat tablets Dosage form: Tablets Specification Appearance: 1.0 mg (pink to pale red) or 5.0 mg/ tablet (yellow) Dosage and Administration: 1 tablet (5 mg/ tablet) once a week, orally administered. Take at least 1 hour before meals or at least 2 hours after meals.
  Combination therapy:
  Fulvestrant injection Dosage form: Injection Appearance: A clear, viscous, colorless to yellowish liquid Specification: 5 ml; 0.25g per vial Dosage and Administration: 500 mg by intramuscular injection. Each 28-day treatment cycle is administered on day 1 and day 15 of the first cycle, followed by day 1 of each subsequent cycle Anlotinib capsules Dosage form: Capsule Appearance: White or off-white powder or granules Dosage and Administration: The recommended dose is 10mg each time, once daily, orally before breakfast. Continuous administration 2 weeks, then 1 week off, that is 3 weeks (21 days) as one course of treatment.
  Interventions: Drug: entinostat; Drug: Fulvestrant; Drug: Anlotinib

INTERVENTIONS:
Drug: entinostat — Entinostat tablets, orally once a week (5 mg); Each treatment cycle lasts for 28 days. Treatment will continue until the subject experiences disease progression, intolerable toxicity, voluntary withdrawal, or any other condition specified in the protocol, whichever occurs first.
Drug: Fulvestrant — Fulvestrant, intramuscular injection, 500 mg each time, administered on d1 and d15 of the first cycle, and on d1 of each subsequent cycle. Each treatment cycle lasts for 28 days. Treatment will continue until the subject experiences disease progression, intolerable toxicity, voluntary withdrawal, or any other condition specified in the protocol, whichever occurs first.
Drug: Anlotinib — Anlotinib, 10mg each time, once daily, orally before breakfast. Take the drug for 2 consecutive weeks and then stop for 1 week, that is, 3 weeks (21 days) as one course of treatment.
  Arms: entinostat + fulvestrant+anlotinib

SUMMARY:
* This study was an open, multicenter phase II clinical trial that enrolled 118 patients with HR+/HER2- with recurrent or progressive advanced breast cancer treated with CDK4/6 inhibitors;
* The study adopted the Simon phase 2 design, and all 20 eligible patients were treated with entinostat + fulvestrant; The study was terminated if no more than 2 patients achieved objective response and continued to enter Phase 2 if no more than 3 patients achieved objective response. In Phase 2, qualified patients were randomly assigned at a ratio of 1:1.5 to either the entestasta + fluvestrus group (Group 1) or the anlotinib + entestasta + fluvestrus group (Group 2), with 39 patients enrolled in group 1 and 59 patients enrolled in group 2; All patients were treated until the subjects' treatment would continue until the subjects experienced disease progression, intolerable toxicity, active withdrawal from treatment, or other conditions specified in the protocol, whichever occurred first.
* During the study period, efficacy evaluations will be conducted every 8 weeks in accordance with the Solid Tumor Efficacy Evaluation Criteria (RECIST) v1.1 until disease progression, the initiation of a new anti-tumor treatment by the subject, or the withdrawal of informed consent, whichever occurs first.
* Continuous safety evaluations will be conducted during the study treatment period. All subjects who have received at least one study treatment will be required to undergo end-of-treatment visits and safety follow-up visits within 7 days and 30±2 days after the last study treatment, respectively.
* The end of the study was defined as the occurrence of disease progression or the end of the study treatment in all subjects, or the early termination of the study for other reasons, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form;
2. Female, aged 18 or above;
3. The patient's Eastern Tumor Collaboration Group (ECOG) physical status is 0-1;
4. The patient's expected survival time is ≥3 months;
5. Breast cancer patients diagnosed as HR-positive and HER-2 negative by tumor histopathological and molecular pathological typing (based on the most recent report); 1) Hormone receptor positive refers to estrogen receptor (ER) positive, progesterone receptor (PR) negative or positive (≥1% positive staining cells are considered receptor positive); 2) HER-2 negative means: the immunohistochemical result of the pathological specimen test is 0 or 1+; Or an immunohistochemical result of 2+ and a negative ISH or FISH test.
6. The subject has received at least one line of endocrine therapy as well as CDK 4/6 inhibitor therapy at an unresectable stage of locally advanced recurrence or metastasis; Or disease recurrence occurred during ET combined with CDK4/6 inhibitors as adjuvant therapy or within 12 months after the end of treatment.
7. The subject has not received chemotherapy or ADC therapy for metastatic disease
8. At least one measurable target lesion was evaluated by the investigator in accordance with RECIST 1.1
9. No known active brain metastases or leptomeningeal disease
10. The patient must have adequate organ function within 1 week (7 days) prior to the initiation of study administration, as defined below:

    * Hematology: Hemoglobin (HgB) ≥80 g/L, platelet count ≥100×109 /L, absolute neutrophil count ≥1.0×10 /L.

Note: Platelet transfusion is not allowed within 3 days before these laboratory tests, red blood cell transfusion is not allowed within 14 days, and hematopoietic growth factor (pegylated G-CSF, 14 days for erythropoietin) is not allowed within 7 days. No blood transfusion or use of auxiliary white blood cell, platelet increase drugs such as cytokines or erythropoietin drugs within 2 weeks prior to the screening test

* Renal function: Serum creatinine (Cre) ≤1.5× upper limit of normal (ULN), or glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2. Urine protein <2+ or 24-hour urine protein quantification <1g
* Liver function: Total bilirubin ≤1.5×ULN; If Gilbert syndrome is present, total bilirubin ≤3 mg/dL; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; If there is liver metastasis, both ALT and AST should be ≤5×ULN; Alkaline phosphatase (ALP) ≤2.5×ULN; If there is bone metastasis, it should be ≤5×ULN.

  9. Echocardiography shows left ejection fraction (LVEF) ≥50% and QTc interval ≤480 ms.

  10. Female patients in the premenopausal or perimenopausal period who agree to use the concomitant luteinizing hormone-releasing hormone (LHRH) agonist can be enrolled. Those who meet any of the following criteria may be considered to have reached menopause, but those who do not meet the criteria for being considered premenopausal or perimenopausal:
* Having undergone bilateral oophorectomy in the past;
* Age ≥60 years;
* Age <60 years old, natural menopause ≥12 months, no chemotherapy, tamoxifen, torremifen or ovarian function castration during this period, blood follicle-stimulating hormone (FSH) and estradiol (E2) levels within postmenopausal range (judged in combination with the reference range of the research center); 11. Patients who are fertile must agree to use recognized effective methods of contraception (including condoms with inactivated sperm, vaginal separators, oral or injectable contraceptives, etc.) or abstain from sexual activity during their participation in the study and for 3 months after the cessation of study treatment.

Exclusion Criteria:

* Patients should not be enrolled if any of the following conditions occur:

  1. Symptomatic visceral metastases or other conditions, visceral crisis, or the investigator deems it inappropriate to use endocrine therapy;
  2. The patient has a past or present central nervous system metastases, or leptomeningeal disease, brain metastases;
  3. Previous use of selective estrogen receptor degraders (SERD, such as fulvestrant) or histone deacetylase (HDAC) inhibitors (such as entectamine, chidamide, etc.) or small molecule multi-target tyrosine kinase inhibitors (such as apatinib, anlotinib, etc.) or PAM pathway inhibitors (such as PI3K inhibitor Alpelisib, AKT inhibitor Capivasertib, MTOR inhibitor everolimus, etc.
  4. Known allergy to SERD, entinostat, or other drugs with a benzamide structure (such as typapride, remopilib, cloprapride, etc.), anlotinib;
  5. Pregnant or lactating women;
  6. Coexisting with other malignant tumors, unless radical treatment has been administered and there is no evidence of recurrence or metastasis;
  7. There is pericardial effusion requiring drainage, pleural effusion with obvious clinical symptoms or ascites;
  8. Other circumstances that the investigator deems unsuitable for inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 118 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-11-25 (Estimated); Study Completion 2028-11-26 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 2 years
  To evaluate the objective response rate (ORR) of entinostat combined with fulvestrant in the treatment of HR+/HER2- advanced breast cancer that has recurred or progressed after CDK4/6 inhibitor therapy.
  Objective response rate was defined as number of patients with complete response (CR) or partial response (PR) divided by all randomized patients. Responses were evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR was defined as disappearance of all target and non-target lesions. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and/or persistence of one or more non-target lesion(s).

SECONDARY OUTCOMES:
PFS | Up to 2 years
  To evaluate progression-free survival (PFS),of entinostat with or without anlotinib + fulvestrant in treatment of relapsed or advanced HR+/HER2- breast cancer treated with CDK4/6 inhibitors
  Progression-free survival (PFS) was defined to be time from randomization to the earliest documented disease progression as defined by the RECIST criteria, new primary breast cancer, or death without progression. The distribution of PFS will be estimated using the Kaplan- Meier method, with 95% confidence intervals calculated using Greenwood's formula. In the primary analysis of PFS, differences in treatment effect will be tested using stratified log rank tests, stratifying on the randomization stratification factors. Stratified univariate and multivariable Cox proportional-hazard models will be built to estimate the hazard ratios (HRs) for treatment effect for PFS as a supportive analysis. In all analyses, P-values will be two-sided.
CBR | up to 2 years
  To evaluate clinical benefit rate (CBR) of entinostat with or without anlotinib + fulvestrant in treatment of relapsed or advanced HR+/HER2- breast cancer treated with CDK4/6 inhibitors
  Percentage of Participants Who Achieve a Best Overall Response of CR, PR or Stable Disease for Greater than or Equal to (≥) 24 Weeks
DoR | Date of CR or PR to date of disease progression or death due to any cause (up to 2 years)
  To evaluate duration of response (DoR) of entinostat with or without anlotinib + fulvestrant in treatment of relapsed or advanced HR+/HER2- breast cancer treated with CDK4/6 inhibitors

OTHER OUTCOMES:
ORR of anlotinib+entinostat+fulvestrant | Up to 2 years
  The objective response rate(ORR) of entesustat combined with anlotinib + fulvestrant in treatment of recurrent or progressive HR+/HER2- advanced breast cancer treated with CDK4/6 inhibitors
  Percentage of Participants Who Achieve a Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Zhejiang, Hangzhou, China